CLINICAL TRIAL: NCT00972036
Title: Phase I Study of Selective Internal Radiation Therapy (SIRT) in Patients With Unresectable Colorectal Cancer Liver Metastases Who Failed Prior Intraarterial Pump Chemotherapy
Brief Title: Selective Internal Radiation Therapy (SIRT) in Patients With Unresectable Colorectal Cancer Liver Metastases Who Failed Prior Intraarterial Pump Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-030
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: COLON; LIVER; RECTUM; SIR-Spheres; 09-030
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unresectable colon cancer patients with liver metastases (Experimental): This study will be performed to evaluate the safety of Selective Internal Radiation Therapy (SIRT) in patients with liver only colorectal cancer metastases that have received hepatic arterial infusion pump and have progressed through at least one line of chemotherapy.
  Interventions: Device: SIR-spheres® (Selective Internal Radiation Therapy)

INTERVENTIONS:
Device: SIR-spheres® (Selective Internal Radiation Therapy) — SIR-spheres® will be administered at 70%, 85% and 100% of the calculated individual patient dose (approximately 1 month prior to SIR-spheres® administration).The first cohort will receive SIRSpheres® at 70% of the individually calculated patient dose, the second will receive 85% of the calculated patient dose, and the third will receive 100% of the calculated patient dose.

SUMMARY:
This study is being done with a new therapy called "Selective Internal Radiation Therapy" (known as SIRT). Radiation is an effective treatment for destroying tumors. It is widely used in cancer treatment. However, radiation can harm normal tissue. SIR-Spheres are tiny plastic beads. They contain a radioactive agent called Yttrium-90. These beads can be delivered through a small tube inserted into the blood vessel that goes directly to the tumor. The radiation goes directly to the tumor. This spares healthy parts of your liver.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of colorectal cancer.
* Unequivocal imaging of hepatic metastases.
* Dominant Liver metastases. (Small amount extrahepatic disease allowed.)
* Unresectable liver metastases.
* Liver Metastases non-eligible for, or progressed after ablation
* Failed prior HAC.
* ECOG performance status 0 - 1
* WBC > or = to 1.5 x 109/L
* Platelets > or = to 50 x 109/L
* Creatinine ≤ 1.5 mg/dl
* Bilirubin ≤ 1.5 mg/dl
* Age > or = to 18 years
* Female patients must either be postmenopausal, sterile (surgically or radiation- or chemically-induced), or if sexually active, must agree to use an acceptable method of contraception.
* Male patients must be surgically sterile, or if sexually active, must agree to use an acceptable method of contraception.
* Life expectancy of at least 3 months without any active treatment.
* No chemotherapy regimen administration for at least 4 weeks prior to SIRT administration

Exclusion Criteria:

* Evidence of severe cirrhosis (CHILDS B and C), portal hypertension with gastroesophageal varices and liver failure as determined by clinical, radiologic or laboratory assessment.
* Previous radiotherapy delivered to the liver.
* Pregnant or breast-feeding.
* Any of the following are contraindications to the use of Yttrium-90 microspheres, and are therefore exclusion criteria:

  * With a Tc-99m macroaggregated albumin (MAA) hepatic arterial perfusion scintigraphy that shows any disposition to the gastrointestinal tract that cannot be corrected by angiographic and embolization techniques.
  * With more than 20% shunting of blood to the lungs as estimated in the Lung Scintigram performed after the intraarterial injection of Tc MAA. Radiation pneumonitis has been seen in patients receiving doses of Yttrium-90 greater than 30 Gy in a single treatment. This corresponds to the shunt over 20% presence of vascular abnormalities, bleeding diathesis, making catheterization of the hepatic artery contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety, toxicity, and maximum tolerated dose of SIR-Spheres® in patients with unresectable metastatic colorectal cancer to the liver (CLM) who have received previous hepatic arterial infusion chemotherapy (HAC). | 2 years

SECONDARY OUTCOMES:
To obtain preliminary evidence of any clinical efficacy of the SIRT therapy in these heavily pretreated patients with unresectable CLM who have received hepatic arterial infusion pump and have failed at least one line of prior chemotherapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Sofocleous, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center 1275 York Avenue, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org